CLINICAL TRIAL: NCT04251208
Title: MOms in REcovery (MORE): Defining Optimal Care for Pregnant Women and Infants
Brief Title: MOms in REcovery (MORE) Study: Defining Optimal Care
Acronym: MORE
Status: Completed | Type: Observational
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sarah E. Lord, Associate Professor of Psychiatry, Biomedical Data Science and Pediatrics; Director, Dissemination and Implementation Core, Center for Technology and Behavioral Health, Trustees of Dartmouth College
Other Study IDs: 00031444
Record Dates: First submitted 2018-11-30; First posted 2020-01-31 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Opioid-Related Disorders; NAS; Substance Use Disorders
Keywords: Pregnancy; Infant, Newborn; Buprenorphine; Methadone; Opiate Substitution Treatment; Comparative Effectiveness; Integrated Care; Referral-based Care; Postpartum; Mental health
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Psychological Well-Being | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrated Care: This is an observational study and no intervention will be administered. The Integrated Cohort consists of pregnant women with identified opioid use disorder who are receiving prenatal care in a maternity setting that provides medication assisted treatment for opioid use.
  Interventions: Other: Observational Study
- Referral-Based Care: This is an observational study and no intervention will be administered. The Referral-Based Cohort consists of pregnant women with identified opioid use disorder who are receiving prenatal care in a maternity setting and are referred to substance use treatment at a specialty care setting.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — No intervention will be administered.

SUMMARY:
Northern New England has among the highest rates of opioid dependence in the U.S, with prevalence highest and growing among those of between the ages of 18-35 years. This region also has among the highest rates of opioid-related deaths in the U.S., with a disproportionate high rate among pregnant women with opioid use disorder. In northern New England (Maine, New Hampshire, & Vermont), 5-8% of newborns have mothers with an opioid use disorder (OUD), greatly increasing the risk of poor outcomes, including preterm birth and long hospitalization for neonatal withdrawal and other newborn complications. For pregnant women with OUD, medication assisted treatment (MAT) significantly reduces these risks. However, it is sometimes difficult for pregnant women to find MAT providers. As a result, many maternity care providers have begun to prescribe MAT in their own practices. Other practices have maintained the longstanding evidence-based standard of care, referral of patients with OUD to specialty MAT treatment program. Most pregnant women with OUD have other psychosocial needs, ranging from lack of housing and untreated mental health conditions, to need for parenting education and support. There is variability among practices in terms of types of other services provided to patients, whether the practice has integrated MAT or relies on referral. Although pregnancy is a time when women are highly motivated to start MAT, many women are also likely to discontinue MAT postpartum due to loss of insurance coverage, difficulty transitioning to another provider, loss of motivation for treatment, or competing demands on time and resources as a new parent.

The challenge for patients, providers, and other stakeholders is to understand the relative advantage of the two MAT models (receiving MAT as part of maternity care or at a specialty program) for improving key outcomes for baby & mother. A second challenge is to understand the relative contributions of onsite services such as mental health care, care coordination, & parenting education to improved outcomes. This question is important to patients & families who may have a choice of where they receive their maternity care. It is even more important in rural areas, such as northern New England, where obstetric practices & specialty care services are limited. Patients, providers & other stakeholders need guidance in choosing the optimal models for building new programs to provide maternity care for women with OUD.

DETAILED DESCRIPTION:
Northern New England has among the highest rates of opioid dependence in the U.S, with prevalence highest and growing among those aged 18-35 years. Regional rates of perinatal opioid use disorders (OUD) reflect this public health crisis; Northern New England region has the highest incidence of opioid-related births in the nation. Perinatal opioid use disorders impact 5-8% of pregnancies in Maine, New Hampshire, and Vermont, three states that have been severely impacted by the current opioid epidemic. Consequences of inadequately treated OUD include premature delivery and other perinatal complications, prolonged newborn hospitalization for neonatal abstinence (NAS), and maternal morbidity and mortality from infectious disease and overdose. In 2013, costs associated with NAS treatment in the U.S. reached $1.5 billion. The epidemic has grown multifold since 2013.

Medication assisted treatment (MAT) with either methadone or buprenorphine is the recommended standard of care during pregnancy. Professionals, including the American College of Obstetricians and Gynecologists (ACOG), the American Academy of Pediatrics, the Society for Maternal-Fetal Medicine, and the American Society for Addiction Medicine, have called to adopt care models that promote early identification and treatment for pregnant women with OUD. Referral to specialty programs for MAT has been the accepted standard of care, with demonstrated safety for women and their infants. However, in response to the escalating opioid crisis, the ACOG began offering buprenorphine training programs to its members. Consequently, a number of maternity care practices throughout Northern New England now provide integrated MAT services. But even where such integrated programs exist, questions persist on the optimal care model for providing MAT to pregnant women with OUD.

There are patient- and provider- factors associated with variability in effectiveness of what MAT model works best for whom. For women, advantages of buprenorphine over methadone include a lower risk of overdose, fewer drug interactions, the accessibility of office-based treatment delivery in the context of maternity care and demonstrated shorter NAS course. The disadvantages of buprenorphine relative to methadone include potential hepatic dysfunction, lack of long-term data on consequences of fetal exposure for infants, potential limited efficacy in patients with high addiction severity, requirement of moderate withdrawal symptoms prior to initiation to avoid iatrogenic withdrawal, and an increased risk of diversion (i.e., sharing or sale). Despite buprenorphine's demonstrated neonatal advantages, it is not effective for all women. The structure of methadone treatment (daily meeting) may also better align with support needs for some women. For providers, the choice of what medication-assisted approach to offer to patients is often restricted by availability and access to specialty care services.

There is limited literature comparing the effectiveness of integrated versus referral MAT care models for postpartum retention in treatment and women's experiences in these two models. In particular, women with high levels of addiction severity or co-occurring mental health conditions may have prenatal care needs from women with less complex behavioral health concerns. Studies have also not assessed the impact of maternal opioid addiction severity on newborn outcomes and maternal long-term recovery. The best neonatal outcomes will be achieved by providing the most appropriate and effective treatment for mothers.

The challenge for patients, providers, and other stakeholders is determining the optimal approach for delivering MAT during pregnancy and after delivery to improve outcomes. Currently, regional obstetrical practices provide either: (1) Integrated care, in which MAT and associated psychosocial services are delivered on site with obstetrical care, and (2) Referral-based care, in which women receive MAT and obstetrical care in separate, specialized locations. Both models have different potential advantages and disadvantages for mothers with OUD and their babies regarding access, availability, acceptability and quality of MAT, obstetrics and other needed services, and long term follow up and treatment after delivery. While pregnancy motivates women to initiate MAT, relapse to use of opioids and cessation of MAT frequently occur during the first postpartum year, placing both mother and infant at significant risk. Payers and policymakers are also seeking answers about where to invest healthcare resources to increase access to treatment for pregnant women, especially in the current opioid crisis. A disproportionate number of women with OUD are insured through the Medicaid system; Medicaid policy affects women's access to a wide range of services, from reimbursement for same-day services or care coordination, to whether a woman continues to be eligible for benefits after delivery.

Study Aims: This study aims to answer these important patient, provider, and policy questions by comparing the real-world effectiveness of two models of MAT delivery currently in clinical use in Maine, New Hampshire, and Vermont with respect to patient experience of care and perinatal, neonatal, and longer-term substance use treatment outcomes.

Two main Comparative Effectiveness Research (CER) Patient-Centered Outcomes Research Institute (PCORI) priority questions will be addressed:

1. Do clinical and patient-reported outcomes for pregnant and parenting women differ between integrated and referral-based MAT practice models?
2. Within models, which psychosocial services are most associated with MAT continuation, and for which groups of patients?

To answer these questions, the following specific aims will be addressed:

Aim 1 (Clinical Outcomes). To use clinical record data to evaluate the comparative effectiveness of Integrated and Referral-Based MAT care models on maternal and neonatal outcomes.

Aim 2 (Patient-reported Outcomes). To use patient reported data to evaluate the comparative effectiveness of Integrated and Referral -Based care models on patient-centered outcomes.

Aim 3 (Heterogeneity of Effects). To examine differences in treatment retention within condition by subgroups of patients based on (1) psychiatric comorbidity, (2) type of medication used for MAT and (3) addiction severity.

Aim 4 (Specification of Services). To determine which services (psychosocial services, care coordination, parenting education) are associated with better maternal and neonatal outcomes.

Aim 5 (Provider). To explore how provider attitudes about MAT and care of patients with OUD vary by care model and are associated with maternal outcomes.

Study Description: This study will collaboratively engage 21 practices providing maternity care across Northern New England, with examples of both integrated care and referral-based models. The study population is pregnant women who receive prenatal care from any of these practices and who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for an opioid use disorder. A cluster-based, prospective observational mixed-methods design will be used to compare outcomes for pregnant women with opioid use disorder receiving prenatal care in obstetric practices that offer MAT through one of two delivery models: Integrated or Referral-based. Clinical records data (n=2000) from pregnant women with OUD receiving prenatal care at a partner practice will be used to examine Aim 1. Aim 2 will be addressed with a patient-report subsample cohort (n=532) recruited in the 3rd trimester of care and followed to 6 months postpartum. Aim 3 will use both kinds of data to explore heterogeneity of treatment effects. For Aim 4, practice-level data will be collected yearly to evaluate services provided across Integrated and Referral-based practices. In Aim 5, survey and qualitative interviews with providers will lend perspective on facilitators and barriers to MAT in both Integrated and Referral-based practice settings. The analytic strategy will account for clustering and patient baseline differences to compare outcomes across assessment points. Whether the effect of treatment type differs according to psychiatric status, type of MAT patients access, or addiction severity will also be tested. Analysis of qualitative data will inform our interpretation of quantitative results and enhance our understanding of patient experience, as well as barriers and facilitators to receiving care within these care models. Patient representatives, practice-partners, state and regional stakeholders, and scientific advisors will actively guide all stages of this study and dissemination of results to relevant partner networks.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 year and older,
* Identified opioid use disorder,
* Receiving prenatal care for current pregnancy at partner practice,
* Clinic-recorded diagnosis of opioid use disorder,
* Willing and able to provide informed consent.

Exclusion Criteria:

* Ward of the State

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Participants will be recruited from our 21 partner maternity care practices located throughout our northeastern New England region: New Hampshire, Maine, and Vermont.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Urine opioid toxicology laboratory report, included in maternal clinical record | Comparison of results at three time points: between 28-36 weeks of pregnancy (third trimester); 36-41 weeks of pregnancy (delivery episode); and at the last documented outpatient postpartum visit (occurring 2-6 weeks after delivery).
  Each clinical record describes the care of the patient over the course of her pregnancy. Urine opioid toxicology results will be reviewed in laboratory reports from each of three time periods. Data collection will include the presence/absence of nonprescribed opioids or metabolites during that time period and measure tracks the change in illicit opioid use across three time periods. Time periods include: third trimester (between 28-36 weeks of pregnancy); delivery episode (between 36-41 weeks of pregnancy); and at the last outpatient postpartum visit (occurring 2-6 weeks after delivery).
Presence or absence of MAT medication in medication list, outpatient narrative, or hospital admission notes included in clinical record. | Comparison of results at three time points: between 28-36 weeks of pregnancy (third trimester); 36-41 weeks of pregnancy (delivery episode); and at the last documented outpatient postpartum visit (occurring 2-6 weeks after delivery).
  Measure is designed to track change in MAT treatment participation by tracking MAT medication use across three time periods- pregnancy, delivery, and postpartum. MAT treatment medications include: buprenorphine, buprenorphine/naloxone, methadone, naltrexone.
Presence or absence of pre-specified perinatal complications in problem list, narrative notes, admission notes in clinical record (Present/Not present). | at time of delivery
  Pre-specified perinatal complications include the following: Hyperemesis, pre-eclampsia, gestational diabetes, prenatal diagnosis of fetal growth restriction, miscarriage, fetal demise, second or third trimester bleeding, placental abruption, maternal mortality, or severe maternal morbidity indicators as defined by CDC: https://www.cdc.gov/reproductivehealth/maternalinfanthealth/smm/severe-morbidity-ICD.htm
Self report (Y/N) of medication assisted treatment (MAT) for opioid use disorder | Comparison of results at three time points: between 28-36 weeks of pregnancy (third trimester); 3 months after delivery, and 6 months after delivery.
  Participant self-report (yes/no) of receiving MAT medicine for opioid use disorder.
Self report on Edinburgh Postnatal Depression Scale (EPDS) (scale) | Comparison of numeric scores at three time points: between 28-36 weeks of pregnancy (third trimester); 3 months after delivery, and 6 months after delivery.
  * Full unabbreviated scale name: Edinburgh Postnatal Depression Scale
  * Maximum and minimum scores: 0-30, higher indicates more severe symptoms
  * Scoring and interpretation of values: A cumulative score of > 10 on the EPDS or any response > 0 for question 10 is considered positive for serious postnatal depression: https://www.knowppd.com/wp-content/uploads/2019/02/edinburgh-postnatal-depression-scale-en.pdf
Self report on Generalized Anxiety Disorders Scale (GAD-7) (scale) | Comparison of numeric scores at three time points: between 28-36 weeks of pregnancy (third trimester); 3 months after delivery, and 6 months after delivery.
  * Full unabbreviated scale name: Generalized Anxiety Disorders Scale- 7
  * Maximum and minimum scores: 0-21, higher indicates more severe symptoms
  * Scoring and interpretation of values: 7-item scale with each item scored from 0 (not at all) to 3 (nearly every day), results are summed to calculate overall score. Score >=10 is considered clinically significant anxiety: https://www.mdcalc.com/gad-7-general-anxiety-disorder-7
Self report on Post-traumatic Stress Disorder Checklist for Civilians (PCL-C) | Comparison of numeric scores at three time points: between 28-36 weeks of pregnancy (third trimester); 3 months after delivery, and 6 months after delivery.
  * Full unabbreviated scale name: Post traumatic Stress Disorder Checklist for Civilians (PCL-C)
  * Maximum and minimum scores: 17-85; higher indicates more severe symptoms.
  * Scoring and interpretation of values: Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point (1-5) scale. Responses range from 1 Not at All - 5 Extremely. Scoring consists of adding up all items for a total severity score: https://www.mirecc.va.gov/docs/visn6/3_ptsd_checklist_and_scoring.pdf

SECONDARY OUTCOMES:
Urine drug/alcohol toxicology laboratory or point of care testing report, included in maternal clinical record | Comparison of results at three time points: between 28-36 weeks of pregnancy (third trimester); 36-41 weeks of pregnancy (delivery episode); and at the last documented outpatient postpartum visit (occurring 2-6 weeks after delivery).
  : Each clinical record describes the care of the patient over the course of her pregnancy. Urine toxicology results will be reviewed in laboratory/point of care testing reports from each of three time periods. Data collection will include the presence/absence of nonprescribed drugs, alcohol, or associated metabolites during that time period and measure tracks the change in illicit drug/alcohol use across three time periods. Time periods include: third trimester (between 28-36 weeks of pregnancy); delivery episode (between 36-41 weeks of pregnancy); and at the last outpatient postpartum visit (occurring 2-6 weeks after delivery).
(Present/Not present). Reference to presence or absence of pre-specified neonatal complications in narrative notes, admission notes in clinical record. | at time of delivery
  Pre-specified neonatal complications include the following conditions: respiratory compromise; infection; neonatal malformation.
Reference to presence or absence of pre-specified neonatal complications in outpatient narrative notes in clinical record (Present/Not present). | at maternal postpartum outpatient visit
  Pre-specified neonatal complications include the following conditions: respiratory compromise; infection; neonatal malformation.
Reference to use of pharmacologic agent to treat neonatal opioid withdrawal in maternal hospital discharge summary or narrative notes (present/absent) | At delivery hospitalization
  The presence or absence of notes indicating the use of one of three medications for pharmacologic treatment for opioid withdrawal in newborns: morphine, methadone, or phenobarbitol
Reference to use of pharmacologic agent to treat neonatal opioid withdrawal in maternal hospital discharge summary or narrative notes (present/absent) | At maternal outpatient postpartum visit
  The presence or absence of notes indicating the use of one of three medications for pharmacologic treatment for opioid withdrawal in newborns: morphine, methadone, or phenobarbitol
Change in Child Custody Status: Self report (Y/N) | compared across two time periods: in the third trimester (between 28-36 weeks of pregnancy); and at 3 and 6 months postpartum
  Retention of child custody (Referral-based practices compared to Integrated care practices; practices with designed care coordinator to practices without designated care coordinator; practices that offer or compared to practices that do not offer psychosocial services; and practices that do not offer parenting education compared to practices that offer parenting education)
Participants recruited through partner maternity care practices and by snowball sampling throughout New Hampshire, Maine, and Vermont. | in the third trimester (between 28-36 weeks of pregnancy)
  Pregnant person age 16 or older Identified diagnosis of OUD Receiving prenatal care for current pregnancy at partner practice Willing and able to provide informed consent
  Exclusion Criteria:
  Under State guardianship, including foster care Incarcerated

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Lord, PhD, Principal Investigator — Dartmouth College; Daisy Goodman, DNP, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (10):
- United States (10):
  - Maine General Hospital, Augusta, Maine
  - Eastern Maine Medical Center/Northern Light, Bangor, Maine
  - Dartmouth Hitchcock Keene/Cheshire Medical Center OB-GYN, Keene, New Hampshire
  - Dartmouth-Hitchcock Medical Center-OB/GYN, Lebanon, New Hampshire
  - Dartmouth Hitchcock Addiction Treatment, Moms in Recovery, Lebanon, New Hampshire
  - Dartmouth Hitchcock Bedford/Manchester, Manchester, New Hampshire
  - Dartmouth Hitchcock Nashua OB-GYN, Nashua, New Hampshire
  - Southwestern Vermont Medical Center OB-GYN, Bennington, Vermont
  - Central Vermont Medical Center, Berlin Corners, Vermont
  - Brattleboro Memorial Hospital OB-GYN, Brattleboro, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko JY, Patrick SW, Tong VT, Patel R, Lind JN, Barfield WD. Incidence of Neonatal Abstinence Syndrome - 28 States, 1999-2013. MMWR Morb Mortal Wkly Rep. 2016 Aug 12;65(31):799-802. doi: 10.15585/mmwr.mm6531a2. PMID 27513154
- [Background] Patrick SW, Schiff DM; COMMITTEE ON SUBSTANCE USE AND PREVENTION. A Public Health Response to Opioid Use in Pregnancy. Pediatrics. 2017 Mar;139(3):e20164070. doi: 10.1542/peds.2016-4070. Epub 2017 Feb 20. PMID 28219965
- [Background] Jones HE. Treating opioid use disorders during pregnancy: historical, current, and future directions. Subst Abus. 2013;34(2):89-91. doi: 10.1080/08897077.2012.752779. PMID 23577898
- [Background] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534
- [Background] Reddy UM, Davis JM, Ren Z, Greene MF; Opioid Use in Pregnancy, Neonatal Abstinence Syndrome, and Childhood Outcomes Workshop Invited Speakers. Opioid Use in Pregnancy, Neonatal Abstinence Syndrome, and Childhood Outcomes: Executive Summary of a Joint Workshop by the Eunice Kennedy Shriver National Institute of Child Health and Human Development, American College of Obstetricians and Gynecologists, American Academy of Pediatrics, Society for Maternal-Fetal Medicine, Centers for Disease Control and Prevention, and the March of Dimes Foundation. Obstet Gynecol. 2017 Jul;130(1):10-28. doi: 10.1097/AOG.0000000000002054. PMID 28594753
- [Background] Jones CM, Campopiano M, Baldwin G, McCance-Katz E. National and State Treatment Need and Capacity for Opioid Agonist Medication-Assisted Treatment. Am J Public Health. 2015 Aug;105(8):e55-63. doi: 10.2105/AJPH.2015.302664. Epub 2015 Jun 11. PMID 26066931
- [Background] Milligan K, Niccols A, Sword W, Thabane L, Henderson J, Smith A, Liu J. Maternal substance use and integrated treatment programs for women with substance abuse issues and their children: a meta-analysis. Subst Abuse Treat Prev Policy. 2010 Sep 1;5:21. doi: 10.1186/1747-597X-5-21. PMID 20809957
- [Background] Wilder C, Lewis D, Winhusen T. Medication assisted treatment discontinuation in pregnant and postpartum women with opioid use disorder. Drug Alcohol Depend. 2015 Apr 1;149:225-31. doi: 10.1016/j.drugalcdep.2015.02.012. Epub 2015 Feb 19. PMID 25735465
- [Background] Flavin J. (2002) A Glass Half Full? Harm reduction amongpregnant women who use cocaine. Journal of Drug Issues, 32(3):973-998. https://journals.sagepub.com/doi/10.1177/002204260203200315
- [Background] Roberts SC, Nuru-Jeter A. Women's perspectives on screening for alcohol and drug use in prenatal care. Womens Health Issues. 2010 May-Jun;20(3):193-200. doi: 10.1016/j.whi.2010.02.003. PMID 20457407
- [Background] Wright TE, Schuetter R, Fombonne E, Stephenson J, Haning WF 3rd. Implementation and evaluation of a harm-reduction model for clinical care of substance using pregnant women. Harm Reduct J. 2012 Jan 19;9:5. doi: 10.1186/1477-7517-9-5. PMID 22260315
- [Background] Jones HE, Heil SH, Baewert A, Arria AM, Kaltenbach K, Martin PR, Coyle MG, Selby P, Stine SM, Fischer G. Buprenorphine treatment of opioid-dependent pregnant women: a comprehensive review. Addiction. 2012 Nov;107 Suppl 1(0 1):5-27. doi: 10.1111/j.1360-0443.2012.04035.x. PMID 23106923
- [Background] Roberts SC, Pies C. Complex calculations: how drug use during pregnancy becomes a barrier to prenatal care. Matern Child Health J. 2011 Apr;15(3):333-41. doi: 10.1007/s10995-010-0594-7. PMID 20232126
- [Background] Terplan M, Kennedy-Hendricks A, Chisolm MS. Prenatal Substance Use: Exploring Assumptions of Maternal Unfitness. Subst Abuse. 2015 Sep 20;9(Suppl 2):1-4. doi: 10.4137/SART.S23328. eCollection 2015. PMID 26448685
- [Background] Thomas CP, Fullerton CA, Kim M, Montejano L, Lyman DR, Dougherty RH, Daniels AS, Ghose SS, Delphin-Rittmon ME. Medication-assisted treatment with buprenorphine: assessing the evidence. Psychiatr Serv. 2014 Feb 1;65(2):158-70. doi: 10.1176/appi.ps.201300256. PMID 24247147
- [Background] Saloner B, Karthikeyan S. Changes in Substance Abuse Treatment Use Among Individuals With Opioid Use Disorders in the United States, 2004-2013. JAMA. 2015 Oct 13;314(14):1515-7. doi: 10.1001/jama.2015.10345. No abstract available. PMID 26462001
- [Background] Fiellin DA, Moore BA, Sullivan LE, Becker WC, Pantalon MV, Chawarski MC, Barry DT, O'Connor PG, Schottenfeld RS. Long-term treatment with buprenorphine/naloxone in primary care: results at 2-5 years. Am J Addict. 2008 Mar-Apr;17(2):116-20. doi: 10.1080/10550490701860971. PMID 18393054
- [Background] Korthuis PT, McCarty D, Weimer M, Bougatsos C, Blazina I, Zakher B, Grusing S, Devine B, Chou R. Primary Care-Based Models for the Treatment of Opioid Use Disorder: A Scoping Review. Ann Intern Med. 2017 Feb 21;166(4):268-278. doi: 10.7326/M16-2149. Epub 2016 Dec 6. PMID 27919103
- [Background] Boyd SC, Marcellus L. (2007) With child: substance use during pregnancy, a woman-centered approach. Halifax [N.S.]: Fernwood Pub.
- [Background] Hall JL, van Teijlingen ER. A qualitative study of an integrated maternity, drugs and social care service for drug-using women. BMC Pregnancy Childbirth. 2006 Jun 13;6:19. doi: 10.1186/1471-2393-6-19. PMID 16772022
- [Background] Lefebvre L, Midmer D, Boyd JA, Ordean A, Graves L, Kahan M, Pantea L. Participant perception of an integrated program for substance abuse in pregnancy. J Obstet Gynecol Neonatal Nurs. 2010 Jan-Feb;39(1):46-52. doi: 10.1111/j.1552-6909.2009.01083.x. PMID 20409102
- [Background] Corse SJ, McHugh MK, Gordon SM. Enhancing provider effectiveness in treating pregnant women with addictions. J Subst Abuse Treat. 1995 Jan-Feb;12(1):3-12. PMID 7752295
- [Background] Armstrong MA, Gonzales Osejo V, Lieberman L, Carpenter DM, Pantoja PM, Escobar GJ. Perinatal substance abuse intervention in obstetric clinics decreases adverse neonatal outcomes. J Perinatol. 2003 Jan;23(1):3-9. doi: 10.1038/sj.jp.7210847. PMID 12556919
- [Background] Goler NC, Armstrong MA, Taillac CJ, Osejo VM. Substance abuse treatment linked with prenatal visits improves perinatal outcomes: a new standard. J Perinatol. 2008 Sep;28(9):597-603. doi: 10.1038/jp.2008.70. Epub 2008 Jun 26. PMID 18580882
- [Background] Meyer M, Phillips J. Caring for pregnant opioid abusers in Vermont: A potential model for non-urban areas. Prev Med. 2015 Nov;80:18-22. doi: 10.1016/j.ypmed.2015.07.015. Epub 2015 Jul 26. PMID 26212632
- [Background] Ordean A, Kahan M, Graves L, Abrahams R, Boyajian T. Integrated care for pregnant women on methadone maintenance treatment: Canadian primary care cohort study. Can Fam Physician. 2013 Oct;59(10):e462-9. PMID 24130301
- [Background] Jansson LM, Velez ML. Infants of drug-dependent mothers. Pediatr Rev. 2011 Jan;32(1):5-12; quiz 12-3. doi: 10.1542/pir.32-1-5. No abstract available. PMID 21196501
- [Background] Terplan M, Ramanadhan S, Locke A, Longinaker N, Lui S. Psychosocial interventions for pregnant women in outpatient illicit drug treatment programs compared to other interventions. Cochrane Database Syst Rev. 2015 Apr 2;2015(4):CD006037. doi: 10.1002/14651858.CD006037.pub3. PMID 25835053
- [Background] Morgenstern J, Blanchard KA, McCrady BS, McVeigh KH, Morgan TJ, Pandina RJ. Effectiveness of intensive case management for substance-dependent women receiving temporary assistance for needy families. Am J Public Health. 2006 Nov;96(11):2016-23. doi: 10.2105/AJPH.2005.076380. Epub 2006 Oct 3. PMID 17018819
- [Background] Dowdell JA, Fenwick J, Bartu A, Sharp J. Midwives' descriptions of the postnatal experiences of women who use illicit substances: a descriptive study. Midwifery. 2009 Jun;25(3):295-306. doi: 10.1016/j.midw.2007.03.008. Epub 2007 Jul 5. PMID 17614166
- [Background] Tuten M, Jones HE. A partner's drug-using status impacts women's drug treatment outcome. Drug Alcohol Depend. 2003 Jun 5;70(3):327-30. doi: 10.1016/s0376-8716(03)00030-9. PMID 12757970
- [Background] Niccols A, Milligan K, Sword W, Thabane L, Henderson J, Smith A. Integrated programs for mothers with substance abuse issues: A systematic review of studies reporting on parenting outcomes. Harm Reduct J. 2012 Mar 19;9:14. doi: 10.1186/1477-7517-9-14. PMID 22429792
- [Background] Niccols A, Milligan K, Smith A, Sword W, Thabane L, Henderson J. Integrated programs for mothers with substance abuse issues and their children: a systematic review of studies reporting on child outcomes. Child Abuse Negl. 2012 Apr;36(4):308-22. doi: 10.1016/j.chiabu.2011.10.007. Epub 2012 Apr 5. PMID 22483158
- [Background] Back SE, Lawson KM, Singleton LM, Brady KT. Characteristics and correlates of men and women with prescription opioid dependence. Addict Behav. 2011 Aug;36(8):829-34. doi: 10.1016/j.addbeh.2011.03.013. Epub 2011 Mar 25. PMID 21514061
- [Background] Back SE, Payne RL, Wahlquist AH, Carter RE, Stroud Z, Haynes L, Hillhouse M, Brady KT, Ling W. Comparative profiles of men and women with opioid dependence: results from a national multisite effectiveness trial. Am J Drug Alcohol Abuse. 2011 Sep;37(5):313-23. doi: 10.3109/00952990.2011.596982. PMID 21854273
- [Background] Najavits LM, Weiss RD, Shaw SR. The link between substance abuse and posttraumatic stress disorder in women. A research review. Am J Addict. 1997 Fall;6(4):273-83. PMID 9398925
- [Background] Chander G, McCaul ME. Co-occurring psychiatric disorders in women with addictions. Obstet Gynecol Clin North Am. 2003 Sep;30(3):469-81. doi: 10.1016/s0889-8545(03)00079-2. PMID 14664322
- [Background] Dube SR, Felitti VJ, Dong M, Chapman DP, Giles WH, Anda RF. Childhood abuse, neglect, and household dysfunction and the risk of illicit drug use: the adverse childhood experiences study. Pediatrics. 2003 Mar;111(3):564-72. doi: 10.1542/peds.111.3.564. PMID 12612237
- [Background] Heffner JL, Blom TJ, Anthenelli RM. Gender differences in trauma history and symptoms as predictors of relapse to alcohol and drug use. Am J Addict. 2011 Jul-Aug;20(4):307-11. doi: 10.1111/j.1521-0391.2011.00141.x. Epub 2011 May 31. PMID 21679261
- [Background] Seng JS, D'Andrea W, Ford JD. Complex Mental Health Sequelae of Psychological Trauma Among Women in Prenatal Care. Psychol Trauma. 2014 Jan;6(1):41-49. doi: 10.1037/a0031467. PMID 25558308
- [Background] Simpson TL, Miller WR. Concomitance between childhood sexual and physical abuse and substance use problems. A review. Clin Psychol Rev. 2002 Feb;22(1):27-77. doi: 10.1016/s0272-7358(00)00088-x. PMID 11793578
- [Background] Benningfield MM, Arria AM, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Fischer G, Jones HE, Martin PR. Co-occurring psychiatric symptoms are associated with increased psychological, social, and medical impairment in opioid dependent pregnant women. Am J Addict. 2010 Sep-Oct;19(5):416-21. doi: 10.1111/j.1521-0391.2010.00064.x. PMID 20716304
- [Background] Jones HE, Svikis D, Rosado J, Tuten M, Kulstad JL. What if they do not want treatment?: lessons learned from intervention studies of non-treatment-seeking, drug-using pregnant women. Am J Addict. 2004 Jul-Sep;13(4):342-57. doi: 10.1080/10550490490483008. PMID 15370933
- [Background] Thompson MP, Kingree JB. The frequency and impact of violent trauma among pregnant substance abusers. Addict Behav. 1998 Mar-Apr;23(2):257-62. doi: 10.1016/s0306-4603(97)00032-4. PMID 9573429
- [Background] Fitzsimons HE, Tuten M, Vaidya V, Jones HE. Mood disorders affect drug treatment success of drug-dependent pregnant women. J Subst Abuse Treat. 2007 Jan;32(1):19-25. doi: 10.1016/j.jsat.2006.06.015. Epub 2006 Oct 13. PMID 17175395
- [Background] Tuten M, Heil SH, O'Grady KE, Fitzsimons H, Chisolm MS, Jones HE. The impact of mood disorders on the delivery and neonatal outcomes of methadone-maintained pregnant patients. Am J Drug Alcohol Abuse. 2009;35(5):358-63. doi: 10.1080/00952990903108231. PMID 20180664
- [Background] Benningfield MM, Dietrich MS, Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Fischer G, Martin PR. Opioid dependence during pregnancy: relationships of anxiety and depression symptoms to treatment outcomes. Addiction. 2012 Nov;107 Suppl 1(0 1):74-82. doi: 10.1111/j.1360-0443.2012.04041.x. PMID 23106929
- [Background] Ashley OS, Marsden ME, Brady TM. Effectiveness of substance abuse treatment programming for women: a review. Am J Drug Alcohol Abuse. 2003;29(1):19-53. doi: 10.1081/ada-120018838. PMID 12731680
- [Background] Flavin J, Paltrow LM. Punishing pregnant drug-using women: defying law, medicine, and common sense. J Addict Dis. 2010 Apr;29(2):231-44. doi: 10.1080/10550881003684830. PMID 20407979
- [Background] Olsen Y, Sharfstein JM. Confronting the stigma of opioid use disorder--and its treatment. JAMA. 2014 Apr 9;311(14):1393-4. doi: 10.1001/jama.2014.2147. No abstract available. PMID 24577059
- [Background] Schroedel JR, Fiber P. Punitive versus public health oriented responses to drug use by pregnant women. Yale J Health Policy Law Ethics. 2001 Spring;1:217-35. No abstract available. PMID 12669331
- [Background] Jansson LM, Svikis D, Lee J, Paluzzi P, Rutigliano P, Hackerman F. Pregnancy and addiction. A comprehensive care model. J Subst Abuse Treat. 1996 Jul-Aug;13(4):321-9. doi: 10.1016/s0740-5472(96)00070-0. PMID 9076650
- [Background] Shaw MR, Lederhos C, Haberman M, Howell D, Fleming S, Roll J. Nurses' Perceptions of Caring for Childbearing Women who Misuse Opioids. MCN Am J Matern Child Nurs. 2016 Jan-Feb;41(1):37-42. doi: 10.1097/NMC.0000000000000208. PMID 26658534
- [Background] Friedrichs A, Spies M, Harter M, Buchholz A. Patient Preferences and Shared Decision Making in the Treatment of Substance Use Disorders: A Systematic Review of the Literature. PLoS One. 2016 Jan 5;11(1):e0145817. doi: 10.1371/journal.pone.0145817. eCollection 2016. PMID 26731679
- [Background] Brener L, Resnick I, Ellard J, Treloar C, Bryant J. Exploring the role of consumer participation in drug treatment. Drug Alcohol Depend. 2009 Nov 1;105(1-2):172-5. doi: 10.1016/j.drugalcdep.2009.06.016. Epub 2009 Jul 21. PMID 19625143
- [Background] Simpatico TA. Vermont responds to its opioid crisis. Prev Med. 2015 Nov;80:10-1. doi: 10.1016/j.ypmed.2015.04.002. Epub 2015 Apr 11. PMID 25869219
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Jumah NA. Rural, Pregnant, and Opioid Dependent: A Systematic Review. Subst Abuse. 2016 Jun 20;10(Suppl 1):35-41. doi: 10.4137/SART.S34547. eCollection 2016. PMID 27375357
- [Background] Oetzel JG, Zhou C, Duran B, Pearson C, Magarati M, Lucero J, Wallerstein N, Villegas M. Establishing the psychometric properties of constructs in a community-based participatory research conceptual model. Am J Health Promot. 2015 May-Jun;29(5):e188-202. doi: 10.4278/ajhp.130731-QUAN-398. Epub 2014 Apr 10. PMID 24720389
- [Background] Oetzel JG, Villegas M, Zenone H, White Hat ER, Wallerstein N, Duran B. Enhancing stewardship of community-engaged research through governance. Am J Public Health. 2015 Jun;105(6):1161-7. doi: 10.2105/AJPH.2014.302457. Epub 2015 Apr 16. PMID 25880952
- [Background] Wallerstein NB, Duran B. Using community-based participatory research to address health disparities. Health Promot Pract. 2006 Jul;7(3):312-23. doi: 10.1177/1524839906289376. Epub 2006 Jun 7. PMID 16760238
- [Background] Sandoval JA, Lucero J, Oetzel J, Avila M, Belone L, Mau M, Pearson C, Tafoya G, Duran B, Iglesias Rios L, Wallerstein N. Process and outcome constructs for evaluating community-based participatory research projects: a matrix of existing measures. Health Educ Res. 2012 Aug;27(4):680-90. doi: 10.1093/her/cyr087. Epub 2011 Sep 21. PMID 21940460
- [Background] Damschroder LJ, Hagedorn HJ. A guiding framework and approach for implementation research in substance use disorders treatment. Psychol Addict Behav. 2011 Jun;25(2):194-205. doi: 10.1037/a0022284. PMID 21443291
- [Background] Hesselink G, Johnson J, Batalden P, Carlson M, Geense W, Groenewoud S, Jones S, Roy B, Sansone C, Wolf JRLM, Bart B, Wollersheim H. 'Reframing Healthcare Services through the Lens of Co-Production' (RheLaunCh): a study protocol for a mixed methods evaluation of mechanisms by which healthcare and social services impact the health and well-being of patients with COPD and CHF in the USA and The Netherlands. BMJ Open. 2017 Sep 7;7(9):e017292. doi: 10.1136/bmjopen-2017-017292. PMID 28882923
- [Background] Portela MC, Pronovost PJ, Woodcock T, Carter P, Dixon-Woods M. How to study improvement interventions: a brief overview of possible study types. BMJ Qual Saf. 2015 May;24(5):325-36. doi: 10.1136/bmjqs-2014-003620. Epub 2015 Mar 25. PMID 25810415
- [Background] Robins JM, Hernan MA, Brumback B. Marginal structural models and causal inference in epidemiology. Epidemiology. 2000 Sep;11(5):550-60. doi: 10.1097/00001648-200009000-00011. PMID 10955408
- [Background] Westfall PH, Tobias RD, Wolfinger RD. Multiple comparisons and multiple tests using SAS. Cary, N.C.: SAS Pub.; 2011
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Stuart EA, Marcus SM, Horvitz-Lennon MV, Gibbons RD, Normand SL. Using Non-experimental Data to Estimate Treatment Effects. Psychiatr Ann. 2009 Jul 1;39(7):41451. doi: 10.3928/00485713-20090625-07. PMID 20563313
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Lee J, Little TD. A practical guide to propensity score analysis for applied clinical research. Behav Res Ther. 2017 Nov;98:76-90. doi: 10.1016/j.brat.2017.01.005. Epub 2017 Jan 19. PMID 28153337
- [Background] Hedeker DR, Gibbons RD. Wiley Series in Probability and Statistics: Longitudinal Data Analysis. 2006. ISBN-13: 978-0471420279
- [Background] Molenberghs G, Kenward MG. Missing Data in Clinical Studies. Chichester: Wiley; 2007. ISBN: 978-0-470-84981-1
- [Background] Varadhan R, Segal JB, Boyd CM, Wu AW, Weiss CO. A framework for the analysis of heterogeneity of treatment effect in patient-centered outcomes research. J Clin Epidemiol. 2013 Aug;66(8):818-25. doi: 10.1016/j.jclinepi.2013.02.009. Epub 2013 May 4. PMID 23651763
- [Background] Lagakos SW. The challenge of subgroup analyses--reporting without distorting. N Engl J Med. 2006 Apr 20;354(16):1667-9. doi: 10.1056/NEJMp068070. No abstract available. PMID 16625007
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Background] Patrick SW, Davis MM, Lehmann CU, Cooper WO. Increasing incidence and geographic distribution of neonatal abstinence syndrome: United States 2009 to 2012. J Perinatol. 2015 Aug;35(8):650-5. doi: 10.1038/jp.2015.36. Epub 2015 Apr 30. PMID 25927272
- [Background] Killip S, Mahfoud Z, Pearce K. What is an intracluster correlation coefficient? Crucial concepts for primary care researchers. Ann Fam Med. 2004 May-Jun;2(3):204-8. doi: 10.1370/afm.141. PMID 15209195
- [Background] McHugo GJ, Drake RE, Whitley R, Bond GR, Campbell K, Rapp CA, Goldman HH, Lutz WJ, Finnerty MT. Fidelity outcomes in the National Implementing Evidence-Based Practices Project. Psychiatr Serv. 2007 Oct;58(10):1279-84. doi: 10.1176/ps.2007.58.10.1279. PMID 17914003
- [Background] Patrick SW, Dudley J, Martin PR, Harrell FE, Warren MD, Hartmann KE, Ely EW, Grijalva CG, Cooper WO. Prescription opioid epidemic and infant outcomes. Pediatrics. 2015 May;135(5):842-50. doi: 10.1542/peds.2014-3299. Epub 2015 Apr 13. PMID 25869370
- [Background] Ordean A, Kahan M, Graves L, Abrahams R, Kim T. Obstetrical and neonatal outcomes of methadone-maintained pregnant women: a canadian multisite cohort study. J Obstet Gynaecol Can. 2015 Mar;37(3):252-257. doi: 10.1016/S1701-2163(15)30311-X. PMID 26001872
- See also: Maine Department of Health and Human Services (DHHS): DHHS to announce the expansion of Medication Assisted Treatment services statewide — http://www.maine.gov/tools/whatsnew/index.php?topic=Portal+News&id=726499&v=article-2016
- See also: American College of Obstetricians and Gynecologists. Medical Education: Responding to a national crisis: Opioid Trainings and Clinical Guidance — https://www.acog.org/About-ACOG/ACOG-Departments/ACOG-Rounds/April-2016/Responding-to-a-National-Crisis-Opioid-Trainings-and-Clinical-Guidance
- See also: Norris L. Maine and Affordable Care Act's (ACA) Medicaid Expansion. 2017 — https://www.healthinsurance.org/maine-medicaid/
- See also: The Henry J. Kaiser Family Foundation. Delivery System Reform Incentive Payment Program (DSRIP) Waivers in Place. 2017 — https://www.kff.org/medicaid/state-indicator/delivery-system-reform-incentive-payment-program-dsrip-waivers-and-uncompensated-care-pools-in-place/?currentTimeframe=0&sortModel=%7B%22colId%22:%22Location%22,%22sort%22:%22asc%22%7D
- See also: Substance Use and Mental Health Services Administration. Behavioral Health Barometer: United States, 2015. Rockville, Maryland: Substance Abuse and Mental Health Services Administration, 2015 — https://www.samhsa.gov/data/sites/default/files/2015_National_Barometer.pdf
- See also: Vandonsel A, Livingston, S., Searle, J. Opioids in Vermont: Prevalence, use, and impact. Vermont Department of Health, 2016 — http://www.healthvermont.gov/sites/default/files/documents/2016/12/ADAP_Opioids_Prevalence_Risk_Impact.pdf
- See also: Maternal Mortality Review Team. Richmond, Virginia: Virginia Department of Health;2015 — http://www.vdh.virginia.gov/content/uploads/sites/18/2016/04/Final-Pregnancy-Associated-Deaths-Due-to-Drug-Overdose.pdf
- See also: American College of Obstetrics and Gynecologists. Statement on Opioid Use During Pregnancy. May 26, 2016 — https://www.acog.org/About-ACOG/News-Room/Statements/2016/ACOG-Statement-on-Opioid-Use-During-Pregnancy
- See also: Substance Use and Mental Health Services Administration. A collaborative approach to the treatment of women with opioid use disorders. Rockville, Maryland: Substance Abuse and Mental Health Services Administration; 2016 — https://ncsacw.samhsa.gov/files/Collaborative_Approach_508.pdf
- See also: World Health Organization Guidelines Review Committee. Guidelines for the identification and management of substance use and substance use disorders in pregnancy. World Health Organization 2014 — https://www.who.int/substance_abuse/publications/pregnancy_guidelines/en/
- See also: The American College of Obstetricians and Gynecologists Statement on Opioid Use During Pregnancy. May 26, 2016 — https://www.acog.org/About-ACOG/News-Room/Statements/2016/ACOG-Statement-on-Opioid-Use-During-Pregnancy?IsMobileSet=false
- See also: Stone R. Pregnant women and substance use: fear, stigma, and barriers to care. Health Justice. 2015;3(1) — https://doi.org/10.1186/s40352-015-0015-5
- See also: Velentgas P, Dreyer NA, Nourjah P, Smith SR, Torchia MM, eds. Developing a Protocol for Observational Comparative Effectiveness Research. Washington, DC: United States Department of Health and Human Services; 2013. AHRQ, ed. — https://www.ncbi.nlm.nih.gov/books/NBK126190/
- See also: SAS Institute Inc. SAS/STAT User's Guide, version 9.4. Cary, NC: SAS Institute Inc.; 2015 — https://www.sas.com/en_us/software/sas9.html
- See also: Patient Centered Outcomes Research Institute Methodology Committee. PCORI Methodology Standards. Washington, DC, 2017 — https://www.pcori.org/research-results/about-our-research/research-methodology/pcori-methodology-standards